CLINICAL TRIAL: NCT04285125
Title: High Resolution Imaging for Analysis of Multinodular and Vacuolating Neuronal Tumor of the Cerebrum
Brief Title: High Resolution Imaging for Analysis of MVNT
Acronym: HAM
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2019_16
Record Dates: First submitted 2019-10-01; First posted 2020-02-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Benign Neuronal Desease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cerebral MRI — Patients who agree to participate in the study will perform an MRI with ultra high resolution sequences added by the research MRI of control will be done at one year and two years

SUMMARY:
MVNT (multinodular and vacuolating neuronal tumor of the cerebrum) is a benign, recently discovered, neuronal lesion, the incidence of which is unknown.

It seems to predominate in the temporal lobes and presents a characteristic MRI appearance: multiple subcortical nodules, developed at the white substance / gray substance junction, of variable size, well limited, in iso-hyposignal T1, hypersignal T2 and hypersignal FLAIR.

The articles describing this entity report the lack of scalability in MRI during patient monitoring, going in the direction of the benignity of the lesion.

The diagnosis sometimes remains uncertain with current MRI sequences, and the patient risks undergoing invasive surgery to remove a lesion that is actually benign. Hence the importance of developing the most precise diagnostic criteria possible. The contribution of advanced MRI techniques, such as ultra-high resolution sequences in the characterization of these lesions, has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Prospective inclusion of all patients with suspected MVNT on a first exploratory MRI: at least the 2 major criteria associated with at least 1 minor criterion will be required to fit into the definition of suspected MVNT:

  * Major criteria :

    * Multinomodular clustered appearance
    * Franc hypersignal FLAIR/T2
  * Minor criteria :

    * No mass effect
    * Hyposignal T1
* Having received informed information about the study and having given express consent to participate in the study

Exclusion Criteria:

* Contraindication to MRI
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Secondary exclusion criteria:

- No characterization MRI done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of MVNT during a first exploratory MRI.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of patients with a central T2 / FLAIR hyposignal visible on standard sequences and on ultra-high resolution sequences. | Day 1
  Among the patients with confirmation of the diagnosis of MVNT (Multinodular and Vacuolating Neuronal Tumor) on the characterization MRI

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Groupe Hospitalier Pellegrin, Bordeaux, Bordeaux
  - CHU Rennes, Rennes, Rennes
  - CHU de Rouen, Rouen, Rouen
  - Hôpital Pierre Paul Riquet, CHU Purpan, Toulouse, Toulouse
  - Fondation A De Rothschild, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Laennec, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No